CLINICAL TRIAL: NCT04301531
Title: Determining the Impact of Scaling up Mass Testing, Treatment and Tracking on Malaria Prevalence Among Children in the Pakro Sub District of Ghana
Brief Title: Determining the Impact of Scaling up Mass Testing, Treatment and Tracking on Malaria Prevalence in Ghana
Acronym: DetI-MTTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: Ghana National Malaria Control Programme (Unknown); Communities (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMIMR
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Malaria Asymptomatic Parasitaemia
Keywords: Malaria; Determine; impact; mass testing and treatment; children under 5; Pakro Ghana
MeSH Terms: conditions — Malaria; Tooth, Impacted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: In the intervention arm, all participants are tested using RDTs and treated if they carry the malaria parasite. This is carried out six times in two years.
  In the control arm participants are only tested and treated if confirmed to be carrying the parasite at baseline and evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (intervention arm) (Experimental): Arm 1 or the intervention arm will involve seven communities: 4-monthly mass screening, and treatment of those who test positive by CHWs will be conducted. Febrile cases will be tested and treated by CHWs any time
  Interventions: Other: Mass testing using RDTs; Drug: Treatment for all cases confirmed positive malaria cases with ACTs; Other: Determination of Hb; Other: Household survey; Other: Community-base management of malaria
- Arm 2 (control arm) (Other): Arm 2 or the Control arm will involve 2 communities: mass screening and treatment only done at baseline and at evaluation. Febrile cases will be tested and treated by CHWs any time.
  Interventions: Other: Mass testing using RDTs; Drug: Treatment for all cases confirmed positive malaria cases with ACTs; Other: Determination of Hb; Other: Household survey; Other: Community-base management of malaria

INTERVENTIONS:
Other: Mass testing using RDTs — To determined the prevalence of asymptomatic malaria parasitaemia. In arm 1 all participants will be tested six times over the study period while in arm 2 the participants will be only be tested at baseline and evaluation.
Drug: Treatment for all cases confirmed positive malaria cases with ACTs — During each mass testing, all confirmed positive cases are treated in both arms.
Other: Determination of Hb — Hb of all children in the subgroup study are measured using a haemocure photometer.
Other: Household survey — Determine the prevalence of febrile illnesses among children in the subgroup study
Other: Community-base management of malaria — Between interventions, participant who become febrile are tested and treated if confirmed positive for malaria by CHWs

SUMMARY:
Globally, malaria prevalence in 2016 was reported to have increased with 445,000 deaths, 91% of which occurred in sub-Sahara Africa with more than 75% being children. Individuals who carry the malaria parasite can either be symptomatic (showing signs and symptoms) or asymptomatic (without signs and symptoms). Asymptomatic malaria parasitaemia pose a very serious threat to malaria control efforts as they serve as reservoirs that fuel the transmission process. Therefore, interventions that target community-wide clearance of asymptomatic parasitaemia can drastically reduce malaria prevalence in the population and lead to elimination especially in endemic areas. Mass parasite clearance can deplete the parasite reservoirs and lower the transmission potential.

Efforts are ongoing to scale-up interventions that work such as use of Long Lasting Insecticidal Nets (LLIN), Intermittent Preventive Treatment in children (IPTc), and test, treat and track (TTT). However, there is need for mass testing, treatment and tracking (MTTT) of the whole population to reduce the parasite load before implementing the aforementioned interventions. Though, Seasonal Malaria Chemoprophylaxis (SMC) is adopted for selected localities in Ghana, the impact of such interventions could be enhanced, if combined with MTTT at baseline to reduce the parasite load. IPT of children in Ghana has demonstrated a parasite load reduction from 25% to 1%. However, unanswered questions include - could this be scaled up? What can be the coverage? What is needed for MTTT scale -up? In a pilot in Ghana, a coverage of more than 75% was achieved in target communities and reduced asymptomatic parasitaemia by 24% from July 2017 to July 2018. It is important to generate time series data to better analyse and understand the prevalence trends as well as the bottlenecks.

In designing interventions that aim at reducing the burden of malaria in children under five, for example, MTTT has largely been left out. This study explores the scale-up of interventions that work using community volunteers, hypothesising that implementing MTTT complemented by community-based management can reduce the prevalence of asymptomatic malaria parasite carriage in endemic communities. The effect of the interventions will be observed by comparing baseline data to evaluation data. This study will document the challenges and bottlenecks associated with scaling-up of MTTT to inform future efforts to scale-up the intervention.

DETAILED DESCRIPTION:
Background Malaria continues to pose a serious burden to the local populations in sub-Sahara Africa. Several efforts have been made to scale up interventions that work such as preventing man-vector contact, intermittent preventive therapy, seasonal malaria chemoprophylaxis as well as TTT for febrile patients. However, much still has to be done to target the mass testing, treatment and tracking of whole populations in order to reduce the parasite load before implementing the above mentioned interventions. Though SMC is adopted for selected localities in Ghana, MTTT could be used to drastically bring down the parasite load in a given population before the implementation of interventions such as SMC. Elsewhere, it has been demonstrated that incorporating the antimalarials in vaccination programmes could delay the first malaria episode in children under five. Furthermore, IPT of children in a community in Ghana has been reported to reduce the parasite load in a given community from 25% to 1%. The questions that remain are - could this be scaled up? What proportion of the community could be covered over a given time? What is needed to accomplish MTTT in large scale? In an ongoing pilot study in Ghana, a coverage of more than 75% was achieved in the target communities and a reduction of 24% in asymptomatic parasitaemia prevalence from July 2017 to July 2018. This proposal is intended to validate the findings of the pilot study.

In designing interventions that aim at reducing the burden of malaria in children under five, e.g, MTTT could be used to clear parasites from the general population before the interventions are implemented. This is because the adults who are not often included in the interventions that target children under 5 years old tend to act as reservoirs that fuel the transmission. To solve the problem of personnel who are limited at the level of the health service and coverage, this study will be making use of the existing network of community health workers (CHWs) that are used during vaccination programmes. The CHWs who reside in the communities, will carry out interventions in their communities and conduct the home-based management of malaria to reduce cost. To solve the problem of stock-outs of RDTs and ACTs, mobile phones SMS will be used. Monthly monitoring and of the volunteers. The volunteers will be trained based on the 2014 Ghana National Malaria Treatment Guidelines for managing uncomplicated malaria.

The study hypotheses that in the Pakro sub district, there are more asymptomatic malaria cases than the symptomatic cases reported by hospital records and that if MTTT is carried out in combination with home-based management of malaria in specific communities over two years, a large proportion of the parasite reservoir will be cleared and consequently open up possibilities for pre-elimination of malaria in the area. It is also intended that the bottlenecks involved in scaling up mass testing, treatment and tracking will be documented in order to facilitate the process.

Over the last decade, the number of recorded malaria cases has steadily dropped from 247 million cases with 881,000 deaths reported in 2006 to 216 million with 445,000 deaths in 2016 (WHO, 2009, 2010, 2016). This has largely been due to the introduction of ACTs following the resistance witnessed against chloroquine as well as an increase in the number of control measures such as the use of long lasting insecticidal nets (LLIN) and intermittent preventive treatment in pregnancy and children. Despite the reported decrease, sub Saharan Africa still bears the greatest burden of the disease where 90% of the deaths are reported with more than 75% of the mortalities in children under five.

Following the recommendation of the WHO, Ghana changed its malaria treatment guidelines adopting artesunate and amodiaquine as first line for the treatment of uncomplicated malaria to replace chloroquine. By 2012, hospital statistics across the country revealed that malaria was responsible for 38.93% of the outpatient consultations and 38.80% of admissions. Studies in Ghana have demonstrated that artesunate and amodiaquine combinations are not only efficacious in clearing the malaria parasites from patients but if used for intermittent preventive treatment for children under five could effectively clear more than 90% of the parasite in this age group.

Different studies have demonstrated very high level of asymptomatic malaria parasitaemia in both less than 5 years old and school age children who have a higher risk of coming down with clinical malaria. The high incidence of asymptomatic parasitaemia serves as a reservoir that fuels the malaria transmission cycle. If the parasite is cleared from the blood of asymptomatic individuals as well as the sick patients with the very efficacious Artemisinin-based Combination Therapy (ACT), then, even the most effective mosquito vector would have nothing to transmit following a blood meal.

As children grow beyond age 5 years, the prevalence of malaria or parasitaemia in this group begins to decrease following the development of immunity to the parasite. A study of trends in malaria admission in Cameroon has demonstrated that the variation in the prevalence of malaria effectively reflected a variation in children age 1 to15 years. While enormous effort is being made to prevent man-vector contact through the use of treated nets, the benefits from using these nets could be amplified if such programmes integrate mass parasite clearance as part of their agenda.

There has been concerted effort in the past decade to evaluate the possible effects of malaria mass treatment using intermittent preventive treatment in under 5 children in different part of Africa. A longitudinal study in Ghana demonstrated that associating IPTc with home based management of malaria by community workers could clear more than 90% of the parasite pool in children using artesunate and amodiaquine. This low level of parasitaemia in the study population was found to persist over a period of two years. Though, this intervention had targeted only under 5 years children, it revealed the potential role intermittent preventive treatment of the population could play in reducing malaria prevalence and consequently paving the way for malaria elimination. Given that old members of the household are likely to have some immunity to the malaria parasite, they however, represent the reservoir that refuels the parasite pool whenever it is reduced by IPTc. Therefore, for intermittent preventive treatment to be sustainable all members of each household should be targeted for mass testing, treatment and tracking and consequent prompt home-based treatment for confirmed cases. Bearing in mind that huge resources are required for IPT of whole communities, it has been suggested that mass screening of whole communities be carried out once a year while IPTc be conducted regularly in combination with the home based management. This could further enhance the efforts.

Implementation of rapid scale-up preventive interventions in the past decade has led to a reasonable decrease in the burden of malaria. The challenges involved with translating research scenarios into implementation are enormous. In an era with a decreased funding for the health system, it is important to understand the bottlenecks that can hinder the scale-up of mass testing and treatment.

This study is aimed at reducing the asymptomatic parasitaemia in the Pakro sub district of Ghana by conducting MTTT for malaria among household members of age 2 months and older and carrying out targeted treatment of all cases with confirmed asymptomatic parasitaemia or clinical malaria. The interventions intend to follow-up an entire population in 24 months.

Main objective:

To determine the impact of scaling up mass testing, treatment and tracking on malaria prevalence among children under fifteen years of age in the Pakro sub district of Ghana.

Specific Objectives:

To assess the effect of scaling-up targeted MTTT/home-based treatment on malaria parasitaemia prevalence.

To determine the prevalence of asymptomatic parasitaemia among afebrile participants <15 years.

To document challenges which hinder the scale up of mass testing, treatment and tracking of malaria in Ghana.

To determine the cost benefit analysis of MTTT to the community

Study Design:

This is a clinical intervention study to be undertaken within a 36 month frame work in 9 communities in the Pakro sub district. The interventions are designed to compare the baseline to evaluation findings following the pilot study. Interventions are determined at the community level. An intervention in this study involves testing the participants with RDTs, the treatment of those who test positive with ACTs and follow up. The study team will undertake 6 household interventions and household surveys over a two-year surveillance period (one intervention/survey every four months). The study will be conducted in two arms - Arm 1 will constitute the intervention communities while Arm 2 will constitute Control Arm communities (standard of care) (Fig 1).

Arm 1 (Intervention arm) will involve seven communities: 4-monthly mass screening, and treatment of those who test positive by CHWs. Febrile cases will be tested and treated by CHWs any time.

Arm 2 (Control arm) will involve 2 communities: mass screening and treatment only done at baseline and at evaluation. Febrile cases will be tested and treated by CHWs any time.

This will allow for the evaluation of the impact of the MTTT without bias in the control Arm. The results from Arm 1 will be compared to Arm 2. Participants in Arm 1 will be tested every four months and treated if positive, while for those in Arm 2, the MTTT exercise will be conducted only at baseline and at evaluation (Fig 1). To avoid the bias that could be introduced by frequent surveys in the control communities with the obligation to treat those that are positive, the number of surveys in Arm 2 are reduced to two - one at baseline and one at evaluation. Those confirmed positive in Arm 2 will be treated and it is believed that this will not affect the study since the baseline and evaluation prevalence data are collected 20 months apart (Fig 2). However, participants in both arms will be monitored by the CHWs - if they become febrile at any time, they will be tested and treated if confirmed positive for malaria. The first intervention is scheduled for month 6 of the grant. Subsequent interventions are scheduled for month 10, 14, 18, 22 and the final intervention is estimated to take place at month 26. CHWs will continue community management of malaria till the 30th month (total study period: 24 months) when the final hospital data will be collected.

In this study a household survey consists of i) measuring the temperature and testing of all participants with RDTs, those who test positive will be treated with ACTs, ii) administration of questionnaires to caregivers to assess the frequency of febrile illnesses and use of mosquito nets in all households and iii) take Hb readings for children <15 years old selected into the study subgroup (see section on participants).

There will be monthly CHW monitoring visits to ensure proper implementation. During each monthly monitoring visit, RDT and ACT stocks will be replenished, and the PI will have a meeting with the CHWs, review what was done and document challenges as well as ensure adherence to SOPs.

Since the study will use RDT for testing, it is known that RDTs do not detect low density infections. This means that there is possibility for transmission to be re-ignited due to low density parasitaemia missed by RDTs (Vásquez, Medina et al. 2018). Despite this flaw, RDTs remain the method of choice to handle large population in a cost effective manner. The challenges faced during implementation will be documented during monitoring. Focus group discussions (FGDs) and in-depth interviews will be organised to obtain additional information from the community and stakeholders such as the NMCP, Regional and District units of the Ghana Health Service and the community. The FGDs and in-depth interviews will be audio taped and the tapes will be store for two years before discarding. Each FDG will last for one hour and involving between 7-15 participants (both men and women). A social scientist and the PI will conducted FDGs and IDI at chosen locations in the communities.

Methodology:

Study Area:

Pakro is one of five sub-districts in the Akwapim south district health directorate (DHD) in the Eastern region of Ghana. The Akwapim south district lies within the semi-equatorial climatic region, and experiences two rainfall seasons in a year, with an average rainfall of 125cm to 200cm. The first rainy season begins from May to June with the heaviest rainfall in June, whilst the second rainy season begins from September to October. According to the Ghana Statistical Service (GSS), the average household size in the Akwapim South district is estimated to be 4.0 whilst the average number of households per house or compound is estimated to be 1.6. The Pakro sub-district has an estimated population of 7,889, and is bounded to the east by Akwapim North district; to the north by Ayensuano district; and to the west by Nsawam Adoagyiri Municipality. The sub-district is made up of 22 communities, and has 3 health care facilities (1 Health Centre and 2 Community-Based Health Planning Service (CHPS) compounds). Due to limited resources, only seven intervention communities will be selected for this study and include Abeasi Newsite, Fante Town, Zongo (Adjenase/Kweitey), Piem/odumsisi, Adesa Latebibio, Sacchi/Tabankro and Odum Tokuro. In consultation with the district health service, all 7 intervention communities which were located within a 5km radius from the health facility were selected. The two control communities (Obosono and Ankwenso) are located out of this zone but are served by two other nearby health facilities. Malaria parasite positivity rate was estimated to be 39.6% in 2014. In the 2014, anaemia among pregnant women at 36 weeks of gestation was 21%.

Study participants:

Community entry activities to sensitise the chiefs and the general population will be conducted at the beginning of the study through meetings. Households will be given unique identification codes. Each individual within the household will be assigned a code that links them to a particular household and community. The intervention will target all the household members. The primary outcome will be based on data from all enrolled under 15 children.The effect of the interventions on secondary outcome 1 will be observed in a subgroup of children aged 2 months to 14 years randomly selected from all the communities in each arm - 460 children in Arm 1 and 395 children in Arm 2. The children in the subgroup will have in addition to the other data, their Hb readings taken to assess the level of Anaemia. The effect of the interventions on secondary outcome 2 will be observed in all under 15 children. Furthermore, the effect of the intervention on secondary outcomes 3 and 4 will be observed in all participants. It is hypothesized that within the study population, the prevalence of asymptomatic parasitaemia should drop by 20% by the end of the first year and by 10% by the end of the second year. In the same light it is expected that anaemia should drop by the same proportion.

Sample size:

This study aims to enrol an entire population estimated at 4500 participants from the 7 selected communities (intervention arm) and the 1500 from two control communities in Pakro sub district. However, to measure the effect of the intervention on secondary outcome such as anaemia in children < 15 years, a sample of 368 children (without correction for loss to follow up) will be needed to determine the malaria prevalence projected at 50% in the study population. This has been determined using the formula of Yamane where n = N/(1+N(e^2)) considering a 95% confident level (CI) and ±5% precision (e). Assuming a loss to follow up of 10% and a non-response rate of 10%, the sample size is readjusted to 460 children calculated from (368/1-0.2) for the community survey. In the control arm, 395 children (316/1-0.2) will be recruited. Questionnaires will be administered to the caregivers of children in the subgroup study. Following a census of the households, children from 2 months to 14 years old will be divided into the various age groups 2 months to 11 months, 1-4 years, 5 -10 years and 11-14 years. From each age group 115 and 99 children will randomly be selected in the intervention and control arms respectively.

Intermittent preventive treatment for the household members. The research team will conduct mass testing (using RDTs) of all children (from 2 months old) and adults residing in the selected communities for the presence of malaria parasites. For this study, the Ag P.f RDT (SD Bioline) which detects histidinie-rich proteins II antigens (HRP-2 Ag) specific to P.falciparum in human blood will be used. The RDTs will be obtained from the Ghana Health service through the NMCP which uses the services of WHO-FIND Lot Testing Programme. To enable follow up studies in a case where treatment failure is reported, 200ul (two drops) of blood will be collected on filter paper. This will be used to determine immunological parameters such as antibody levels to specific antigens using PCR and ELISA. This is however, not part of this study. All participants confirmed for malaria will be treated using ACTs following Guidelines. If a participant vomits within 30 minutes following treatment, it will be repeated.

Follow-Up:

CHWs will treat all positive cases directly using directly observed treatment (DOT). All treated cases will be followed-up by trained CHW on day 1, 2, 3 and 7 post-treatment to document any adverse events.

Questionnaire:

The questionnaire will include questions about malaria treatment, prevention and control measures practiced by the household members as well as the cost of seeking for treatment. In order to determine the perceived benefit of MTTT, data will be collected on the cost of accessing treatment from community members through in-depth interviews and FGDs.

Training of data collectors Two Community Health Workers (CHWs) will be selected from each community and trained. training will focus on national malaria treatment guidelines - testing using RDTs, treatment with ACTs and follow up as well as home-based management of malaria.

Timely treatment of suspected febrile malaria cases in the community:

Between one MTTT intervention and the next, the trained community members will provide prompt home-based treatment for children and adults reporting signs and symptoms of malaria and confirmed to be carrying the parasite using RDTs. There is a need to visit the health facilities that service the community to enable tracking and linking of medical records with study participants. Hypothesis: a reduction in parasite load in the community could lead to a reduction in the number of malaria related consultations.

Data collection:

Following consent, blood will be drawn from a finger prick by trained CHW. All participants will be tested for the presence of malaria parasites using RDTs and positive cases will be treated. All samples will be stored at NMIMR. To test for anaemia in children in the subgroup a portable automated Hemocue photometer will be used to determine the concentration of Haemoglobin. Anaemia in this study is defined as Hb levels less than 10g/dl. Children with severe anaemia (Hb less than 7g/dl) will be referred to the health facility. To determine the cost benefit of the project, data will be collected on the benefits of the project to the community at the level of the household over the project period. This will include the cost saved through averted cases of malaria at the level of the household plus the cost saved from time lost to providing care when a family member is sick of malaria. A household will be said to have benefited from MTTT if it perceives that by participating in the project, a number of malaria cases were adverted for that year. To place value on each malaria case a household perceives to have adverted, cost of accessing treatment will be determined. Data will be collected on cost the family would have incur in managing each malaria case - transportation (C1), consultation (C2), laboratory (C3) and treatment cost (C4) as well as total indirect cost estimated as lost in activity time as a result of caregiving to the malaria patients (C5). The time lost in caregiving will be estimated using the method of Hutton and Haller, 2004. The benefit will be calculated with a 5% interest rate per year for 2 years after project is completes.

Data Management and Analysis:

A database will be created to manage the data. Data will be entered into Epi-info and analysed using SPSS. The unit of enrolment will be the household. The data will be collected first on paper based case report forms (CRF) before being entered into the database. As a quality control measure, every day, all data collected will be cross checked by the research assistant and validated. If data is not validated due to errors or poor recording, a data query sheet is completed and returned to the person involved to rectify the error before work continues the next day. Once the error is rectified the responsible team members signs and forwards the data to the research assistant who validates it. Once validated the data is moved to the statistic unit of NMIMR. The statistician receives the data and cross checks. In case of any queries the data is returned to the field coordinator for rectification. To assure quality, the process will be closely monitored following a monthly schedule. The data is owned by the NMIMR.

Ethical Consideration:

The ethical clearance for this study will be sought from the NMIMR IBR and GHS-ERC

Privacy and confidentiality All information/samples obtained from participants will be kept confidential and will not be released to a third party. This information will be stored in a secure location at the Epidemiology Department of NMIMR.

Safety Consideration:

There are no health threatening risk involved in this study. The table below describes the potential risk and how it will be mitigated within the framework of this study.

Dissemination of results and Publication The study results will be discussed at every stage with stakeholders (Communities, sub district, district and regional offices of GHS, NMCP, WHO country office) and published in open access peer reviewed journals. Data generated from this study will be stored in two secure databases. A database created for this project in the information technology (IT) unit of NMIMR whose password will be known only to the head of the IT unit and the PI. Data resulting from this work will be used in informing the NMCP decision to develop guidelines for implementing MTTT. The impact of this study will be communicated to the public through durbars with the local communities and chiefs, radio/TV talk shows and appropriate use of social media through blogs and twitter.

Statistical Analysis Baseline Comparison of Patients: Summary statistics (proportions for categorical variables, and means or medians with variances or IQRs for continuous variables) and graphs will be used to detect presence of outliers or unusual observations, and to assess validity of assumptions for statistical tests. Participants will be compared between the two study arms (Intervention communities and control communities) with respect to baseline demographic, clinical and parasitological characteristics. Statistical analysis of the above comparisons for continuous variables will be based on graphs, t-test (or Wilcoxon test), and ANOVA (or Kruskal-Wallis test). Categorical variables will be compared using chi-square tests. All analyses will be performed for the whole population in each arm Primary objective: outcomes of primary objective asymptomatic parasitaemia will be compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Adjustments for potential confounders including patient's age and use of ITN and baseline temperature will be considered. In addition, these outcomes will also be compared over time using Cochrane Armitage test of trends.

Secondary objectives: symptomatic parasitaemia at the hospitals and symptomatic parasitaemia picked up at the community compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Comparisons of anaemia in children <15 years across time and study arms will be assessed through Cochrane Armitage test of trends and using chi-square tests (or fisher exact tests) respectively. A binomial logistic regression will be used to test impact of intervention on febrile illnesses.

Data from FGDs and IDI will be analysed using INVIVO ver 12.

The cost benefit analysis will be calculated as follows:

Net Present Value (NPV) = ∑PV of all the Expected Benefits - ∑PV of all the MTTT Associated Costs

Anticipated impact of proposed work

Besides an implementation research, this is also a capacity-development project. The overarching goal of this project is to develop the skills of a multidisciplinary team of researchers and community health workers to improve research through assessing the impact of scaling up MTTT to reduce malaria morbidity and mortality.

It is intended that this project serve as a bench mark for the development of evidence based guidelines for the scale-up of mass testing, treatment and tracking of malaria in sub-Sahara Africa.

Quality Assurance

In order to ensure the quality of data collected, 20 community health workers will be trained and 14 will be selected for the project. The questionnaires will be pretested and corrections effected. All data collected will be cross checked by two persons in the fields. To avoid loss of data, all data from the field will be record in the data transfer sheet be transfer to the data management unit. All ACTs (AL) and RDTs will be procured from the NMCP through the Eastern Region medical store. The expiry dates for all procurements made will be verified.

ELIGIBILITY:
Inclusion Criteria:

1. Overall inclusion criteria for MTTT:

   * Be aged 2 months or older
   * Be resident in the study area
   * Have completed and signed the consent for adults or assent form for children 12-17 years.
2. Inclusion Criteria for children in the subgroup study:

   * Be age range 6 months to 14 years
   * Be resident in the study area for the period of the study.
   * Be willing to participate
   * Parent or guardian have completed and signed consent form
   * Provided assent for children 12-17 years

Exclusion Criteria:

* If an individual intents to stay less than one year in the study site
* Be absent at some time because he/she is schooling in a boarding school
* Has a life threatening illness (excluding malaria).

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5861 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The effect of MTTT/home-base management of malaria on malaria prevalence in children | 2 years
  The difference in asymptomatic malaria parasitaemia prevalence in children <15 years in the intervention arm compared to the control arm.

SECONDARY OUTCOMES:
Prevalence of anaemia in <15 children | 2 years
  The difference in the prevalence of anaemia in children <15 years in the intervention arm compared to the control arm
Prevalence of febrile illnesses | 2 years
  The difference in prevalence of febrile illnesses in children <15 years in the intervention arm compared to the control arm
Prevalence of asymptomatic malaria parasitaemia among household members | 2 years
  The difference in asymptomatic malaria parasitaemia prevalence in household members in the intervention arm compared to the control arm.
Difference in symptomatic malaria cases attending health facilities | 2 years
  The difference in symptomatic malaria cases attending health facilities from households in the intervention arm compared to the control arm.
Cost benefit analaysis of implementing MTTT | 2 years
  The difference in cost benefit of MTTT between arm 1 and arm 2

CONTACTS AND LOCATIONS:
Overall Officials: Ndong Ignatius Cheng, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Noguchi Memorial Institute for Medical Research, Accra, Greater, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahorlu CK, Koram KA, Seake-Kwawu A, Weiss MG. Two-year evaluation of Intermittent Preventive Treatment for Children (IPTc) combined with timely home treatment for malaria control in Ghana. Malar J. 2011 May 15;10:127. doi: 10.1186/1475-2875-10-127. PMID 21569634
- [Background] Bousema T, Okell L, Felger I, Drakeley C. Asymptomatic malaria infections: detectability, transmissibility and public health relevance. Nat Rev Microbiol. 2014 Dec;12(12):833-40. doi: 10.1038/nrmicro3364. Epub 2014 Oct 20. PMID 25329408
- [Background] Bull PC, Lowe BS, Kortok M, Molyneux CS, Newbold CI, Marsh K. Parasite antigens on the infected red cell surface are targets for naturally acquired immunity to malaria. Nat Med. 1998 Mar;4(3):358-60. doi: 10.1038/nm0398-358. PMID 9500614
- [Background] DISTRICT HEALTH DIRECTORATE, 2015. District Annual Report 2015, Akwapim South, Aburi, Ghana
- [Background] Dicko A, Sagara I, Sissoko MS, Guindo O, Diallo AI, Kone M, Toure OB, Sacko M, Doumbo OK. Impact of intermittent preventive treatment with sulphadoxine-pyrimethamine targeting the transmission season on the incidence of clinical malaria in children in Mali. Malar J. 2008 Jul 8;7:123. doi: 10.1186/1475-2875-7-123. PMID 18611271
- [Background] Ansah EK, Narh-Bana S, Affran-Bonful H, Bart-Plange C, Cundill B, Gyapong M, Whitty CJ. The impact of providing rapid diagnostic malaria tests on fever management in the private retail sector in Ghana: a cluster randomized trial. BMJ. 2015 Mar 4;350:h1019. doi: 10.1136/bmj.h1019. PMID 25739769
- [Background] GNMCP 2006. Ghana National Malaria Control Programme: Ghana Health Service Report 2006 Accra.
- [Background] GHANA STATISITCAL SERVICE, 2010. Population and Housing Sensus. District Analytic Report: Akwapim South District.
- [Background] ISRAEL, G. D. 1992. Determining sample size, University of Florida Cooperative Extension Service, Institute of Food and Agriculture Sciences, EDIS.
- [Background] Koram K, Quaye L, Abuaku B. Efficacy of amodiaquine/artesunate combination therapy for uncomplicated malaria in children under five years in ghana. Ghana Med J. 2008 Jun;42(2):55-60. PMID 19180204
- [Background] Kweku M, Webster J, Adjuik M, Abudey S, Greenwood B, Chandramohan D. Options for the delivery of intermittent preventive treatment for malaria to children: a community randomised trial. PLoS One. 2009 Sep 30;4(9):e7256. doi: 10.1371/journal.pone.0007256. PMID 19789648
- [Background] Ndong IC, van Reenen M, Boakye DA, Mbacham WF, Grobler AF. Trends in malaria admissions at the Mbakong Health Centre of the North West Region of Cameroon: a retrospective study. Malar J. 2014 Aug 22;13:328. doi: 10.1186/1475-2875-13-328. PMID 25145498
- [Background] Newell K, Kiggundu V, Ouma J, Baghendage E, Kiwanuka N, Gray R, Serwadda D, Hobbs CV, Healy SA, Quinn TC, Reynolds SJ. Longitudinal household surveillance for malaria in Rakai, Uganda. Malar J. 2016 Feb 9;15:77. doi: 10.1186/s12936-016-1128-6. PMID 26861943
- [Background] Ofosu-Okyere A, Mackinnon MJ, Sowa MP, Koram KA, Nkrumah F, Osei YD, Hill WG, Wilson MD, Arnot DE. Novel Plasmodium falciparum clones and rising clone multiplicities are associated with the increase in malaria morbidity in Ghanaian children during the transition into the high transmission season. Parasitology. 2001 Aug;123(Pt 2):113-23. doi: 10.1017/s0031182001008162. PMID 11510676
- [Background] OTUPIRI, E., YAR, D. & HINDIN, J. 2012. Prevalence of Parasitaemia, Anaemia and treatment outcomes of Malaria among School Children in a Rural Community in Ghana. Journal of Science and Technology (Ghana), 32, 1-10.
- [Background] Rao VB, Schellenberg D, Ghani AC. Overcoming health systems barriers to successful malaria treatment. Trends Parasitol. 2013 Apr;29(4):164-80. doi: 10.1016/j.pt.2013.01.005. Epub 2013 Feb 14. PMID 23415933
- [Background] Sarpong N, Owusu-Dabo E, Kreuels B, Fobil JN, Segbaya S, Amoyaw F, Hahn A, Kruppa T, May J. Prevalence of malaria parasitaemia in school children from two districts of Ghana earmarked for indoor residual spraying: a cross-sectional study. Malar J. 2015 Jun 25;14:260. doi: 10.1186/s12936-015-0772-6. PMID 26109461
- [Background] Sinclair D, Zani B, Donegan S, Olliaro P, Garner P. Artemisinin-based combination therapy for treating uncomplicated malaria. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD007483. doi: 10.1002/14651858.CD007483.pub2. PMID 19588433
- [Background] Farnert A, Snounou G, Rooth I, Bjorkman A. Daily dynamics of Plasmodium falciparum subpopulations in asymptomatic children in a holoendemic area. Am J Trop Med Hyg. 1997 May;56(5):538-47. doi: 10.4269/ajtmh.1997.56.538. PMID 9180605
- [Background] WORLD HEALTH ORGANISATION Roll Back Malaria Report. Geneva: WHO; 2003. http://www.rollbackmalaria.org/microsites/wmd2011/amr_toc.html. Accessed 15 November. 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2009. Geneva: WHO; 2009 http://www.who.int/malaria/world_malaria_report_2014/en. Accessed 3 December. 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2010. Geneva: WHO; 2010. http://www.who.int/malaria/world_malaria_report_2010/en. Accessed 1 December 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2011. Geneva: WHO; 2013 http://www.who.int/malaria/publications/world_malaria_report_2013/en. Accessed 2 December 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2014. Geneva: WHO; 2014 http://www.who.int/malaria/publications/world_malaria_report_2014/en. Accessed 1 December, 2016